CLINICAL TRIAL: NCT06708871
Title: Thermal Ablation Versus Parathyroidectomy for Primary Hyperparathyroidism: a Multicenter Study
Brief Title: Thermal Ablation Versus Parathyroidectomy for Primary Hyperparathyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Other Study IDs: S2024-546-01
Record Dates: First submitted 2024-11-10; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-06

CONDITIONS: Cure Rate; Complication Rate; Efficacy and Safety
MeSH Terms: interventions — Transurethral Resection of Prostate; Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Therma ablation
  Interventions: Procedure: Thermal ablation
- Parathyroidectomy
  Interventions: Procedure: Parathyroidectomy

INTERVENTIONS:
Procedure: Thermal ablation — Thermal ablation is a minimally invasive procedure used to treat primary hyperparathyroidism, a condition where one or more of the parathyroid glands produce excessive amounts of parathyroid hormone (PTH). The treatment involves using heat to destroy the overactive parathyroid tissue. This can be done through various methods such as radiofrequency ablation (RFA) and microwave ablation(MWA).
  Groups: Therma ablation
Procedure: Parathyroidectomy — Parathyroidectomy is a surgical procedure to remove one or more of the parathyroid glands in cases of hyperparathyroidism.
  Groups: Parathyroidectomy

SUMMARY:
This study is a prospective, multicenter study designed to compare the efficacy and safety of surgical treatment versus ablation therapy (including radiofrequency ablation and microwave ablation) for patients with primary hyperparathyroidism (PHPT). The study will assess the impact of both treatment modalities on serum parathyroid hormone (iPTH) and calcium levels, clinical symptom improvement, bone mineral density enhancement, reduction in the incidence of urinary system stones, and postoperative complication rates. While surgical treatment has been the standard of care for PHPT, offering definitive cure, it carries inherent surgical risks and complications. Ablation therapy, as a minimally invasive approach, presents a novel alternative with reduced trauma and fewer complications. The outcomes of this study will inform clinical decision-making and potentially optimize treatment strategies for patients with PHPT.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with primary hyperparathyroidism, such as those with symptoms in any system including the kidneys, bones, gastrointestinal tract, psychoneurological system, or those with atypical symptoms such as muscle weakness, dysfunction, and sleep disorders.
* Asymptomatic PHPT patients with any of the following conditions:

  ① Serum calcium is higher than the upper limit of the normal value by 1 mg/dL (0.25 mmol/L);

  ② There is objective evidence of renal involvement, including asymptomatic kidney stones, nephrocalcinosis, hypercalciuria (24 - hour urinary calcium level > 400 mg/dL) on renal imaging, or impaired renal function (glomerular filtration rate < 60 mL/min);

  ③ There is evidence of osteoporosis (bone mineral density decreased by 2.5 standard deviations at any site) and/or radiographic evidence of fragility fractures.

  ④ Age < 50 years

  ⑤ The patient cannot accept routine follow - up observation.
* Imaging examination shows that at least one parathyroid gland is enlarged.

Exclusion Criteria:

* diagnosis of secondary or tertiary HPT
* severe coagulation disorder
* severe cardiopulmonary insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have a confirmed diagnosis of PHPT based on biochemical and clinical evaluations. Biochemical evidence includes elevated parathyroid hormone (PTH) levels in conjunction with hypercalcemia (serum calcium above the normal reference range). Clinical manifestations may include, but are not limited to, bone pain, osteoporosis, kidney stones, or other symptoms related to the disease.All patients must provide written informed consent after a detailed discussion of the study procedures, potential risks, and benefits of both thermal ablation and surgical treatment options. This ensures that patients are fully aware of what participation in the study entails and have voluntarily agreed to take part.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2024-11-26 (Estimated); Primary Completion 2028-11-26 (Estimated); Study Completion 2028-12-26 (Estimated)

PRIMARY OUTCOMES:
cure rate | 6 months after surgery or ablation
  The cure rate is the probability that postoperative levels of parathyroid hormone (PTH) and blood calcium reach the target values.

SECONDARY OUTCOMES:
complication rate | within 30 days after surgery or ablation
  The incidence rate of complications refers to the proportion of patients who experience complications after a surgical procedure within a certain period.
symptom remission rate | 1 year after treatment initiation
  The symptom remission rate refers to the proportion of the number of patients whose symptoms have been alleviated to the total number of patients treated in the treatment of primary hyperparathyroidism, either by surgery or ablation.
Normalization Probability of Serum Calcium and Phosphorus after Ablation or Surgery | 6 months post-treatment
  The probability of normal serum calcium and serum phosphorus levels after ablation or surgical treatment for primary hyperparathyroidism is defined as the proportion of patients in whom the levels of blood calcium and blood phosphorus return to the normal physiological range among all the patients who have received either ablation or surgical procedures for this condition.
Bone mineral density change | 2 years
  Bone mineral density change after treatment is defined as the alteration in bone density measured by DEXA in patients with primary hyperparathyroidism after surgery or ablation.

OTHER OUTCOMES:
Cosmetology Scoring（Scar Cosmesis Assessment and Rating Scale） | at 3 months, 6 months, and 1 year post-procedure
  The Scar Cosmesis Assessment and Rating Scale (SCAR) will be utilized to evaluate the cosmetic outcome following surgical or ablation treatment for primary hyperparathyroidism. The observer part of the SCAR assesses six aspects: scar spread, erythema, pigmentation abnormality, surgical marks or suture tracks, hypertrophy/atrophy, and overall impression. The patient part includes two simple questions about patient satisfaction with the scar and the degree of itching. The scale has a minimum value of 0, representing the least severe scar with the best cosmetic appearance, and a maximum value of 15, signifying the most severe scar with the poorest cosmetic result. Higher scores on this scale indicate a worse cosmetic outcome.
Readmission Rate within 30 Days | within 30 days after surgery or ablation
All - cause mortality rate | 2 years
Evaluation of the Learning Curve for Surgical and Ablation Procedures in Treating Primary Hyperparathyroidism: Incorporating Key Performance Indicators and Patient Cure Outcomes | through study completion, an average of 2 year
  The learning curve for surgical or ablation procedures will be evaluated by tracking and analyzing key performance indicators, with patient cure outcomes also taken into account. These indicators encompass the time taken from the start of the procedure until its completion (operation time). Additionally, the rate of occurrence of immediate and short-term post-operative complications (like bleeding, nerve injury) is considered. Patient cure status, such as complete remission of related symptoms, normalization of relevant physiological indicators, and long-term disease-free survival, will be meticulously assessed to comprehensively evaluate the effectiveness and learning the effectiveness and learning curve of these procedures.

IPD SHARING:
Plan to Share IPD: No